CLINICAL TRIAL: NCT05565469
Title: Correlation Between Abdominal Wall Stimulation and Neurostimulator Tip Location
Acronym: CAWSAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B2432022000021
Record Dates: First submitted 2022-09-22; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Neurostimulator; Complication; Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neurostimulator group (Experimental): Adjustment of neurostimulator settings to see whether or not abdominal stimulation can be provoked
  Interventions: Other: Adjustment of neurostimulator settings

INTERVENTIONS:
Other: Adjustment of neurostimulator settings — This is an interventional prospective study. After obtaining informed consent, only necessary information will be extracted through the electronic patient record. Through post-operative imaging, a level determination of the neurostimulator tip will be done. During general consultations, patients will be asked if they experienced abdominal wall stimulation after the procedure and when (YES/NO, NRS). This will include looking at the settings of the neurostimulator. And its adjustments. Furthermore, general epidemiological characteristics such as age, gender, height, weight will be extracted from the electronic patient record.
  At the consultation, another active programming will take place (in accordance with clinical programming) on the tip of the electrode to check whether it provokes abdominal wall stimulation. This will also be scored YES/NO + NRS. Then the settings will be returned as they were pre-consultation.

SUMMARY:
In this prospective interventional study, we look at the level of tip of the DTM neurostimulator and the presence of abdominal wall stimulation in patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with a DTM neurostimulator for Failed Back Surgery Syndrome (FBSS) at the thoracic level

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients who are not able to exercise their will.
* Inability to understand the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-23 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-27 (Estimated)

PRIMARY OUTCOMES:
Abdominal stimulation | up to 15 minutes after start of the intervention
  Is abdominal wall stimulation present YES/NO and if so what is the score between 0 and 10 on an NRS 1-10. This is then correlated to the position of the electrode.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Plazier, dr., Principal Investigator — Jessa Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vanloon M, Raymaekers V, Meeuws S, de Ridder D, Plazier M. Correlation Between Abdominal Wall Stimulation and Spinal Cord Stimulator Tip Location: A Nonrandomized Clinical Trial. Neuromodulation. 2023 Oct;26(7):1459-1464. doi: 10.1016/j.neurom.2023.07.004. Epub 2023 Aug 23. PMID 37632515